CLINICAL TRIAL: NCT05901740
Title: Prevalence of Fuctional Heartburn in Patients With IBS .
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed fawzy, Resident, Assiut University
Other Study IDs: Heart burn in IBS Patients
Record Dates: First submitted 2023-06-05; First posted 2023-06-13 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Heartburn
MeSH Terms: conditions — Heartburn

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to assess prevalence of functional heartburn in IBS patients.

DETAILED DESCRIPTION:
Functional heartburn (FH) and IBS are functional digestive disorders that may occur in the same patients (1).

Heartburn is a burning sensation in the chest, radiating toward the mouth, as a result of acid reflux into the esophagus. However, only a small percentage of reflux events are symptomatic. Heartburn is also often associated with a sour taste in the back of the mouth with or without regurgitation of the refluxate.(2) Definition of FH has been greatly modified from the Rome II criteria (in which the definition of FH included all NERD patients with negative pH-manometry) to the Rome III criteria (in which FH is defined as a functional esophageal disorder unrelated to GERD and characterized by negative pH-manometry, the lack of a relationship between symptoms and reflux events, and the lack of symptom improvement after a trial of PPI therapy)(2).

However, data establishing a solid link between FH and IBS are lacking, because the clinical definition of FH has undergone substantial changes over the years(3). the prevalence of IBS varied from 5 to 65% and the incidence varied from 1 to 36% , Its frequency in women is more than men.(4). Psychological problems were strongly associated with prevalence and incidence of IBS. (5) Distinguishing between irritable bowel syndrome (IBS) and functional dyspepsia can be challenging because of the variations in symptom patterns, which commonly overlap.(6) Currently, The criteria for diagnosis of Functional heartburn (FH) rest not only on compatible symptoms but also on exclusion of structural and metabolic disorders that might mimic the functional disorders, Patients have to have a normal X_ray ,normal upper endoscopy and 24-hour PH monitoring test that is normal, and the absence of any evidence of a correlation between physiologic reflux events, either weakly acidic or acidic, and heartburn symptoms.(7,8)

ELIGIBILITY:
Inclusion Criteria:

1. Age above 18 years.
2. Patients diagonsed as IBS (according to the Rome criteria of the lV revision) and presented with heartburn with a normal X_ray, normal upper endoscopy and normal 24-hour PH monitoring.

Exclusion Criteria:

1. Patients who refuse to contribute in this study.
2. Presence of duodenal or gastric ulcer or cancer on upper endoscopy.
3. cardiac patients.
4. Pregnancy and breastfeeding

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The Data will be collected by a questionnaire includes the many dimensions ,one of the most important dimensions is symptoms, including typical and atypical symptoms of GERD. Another assessment dimension is the response to treatment, in which the change in severity and/or frequency of symptoms is measured. A third assessment dimension is diagnosis, a tool to discriminate patients with GERD from other diseases. Also, disease-specific quality of life, the burden of GERD on the quality of life of patients, is an assessment dimension of GERD.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
The purpose of this study is to assess prevalence of functional heartburn in IBS patients. | Baseline
  , The criteria for diagnosis of Functional heartburn (FH) rest not only on compatible symptoms but also on exclusion of structural and metabolic disorders that might mimic the functional disorders, Patients have to have a normal X_ray ,normal upper endoscopy and 24-hour PH monitoring test that is normal, and the absence of any evidence of a correlation between physiologic reflux events, either weakly acidic or acidic, and heartburn symptoms

REFERENCES:
- [Background] de Bortoli N, Martinucci I, Bellini M, Savarino E, Savarino V, Blandizzi C, Marchi S. Overlap of functional heartburn and gastroesophageal reflux disease with irritable bowel syndrome. World J Gastroenterol. 2013 Sep 21;19(35):5787-97. doi: 10.3748/wjg.v19.i35.5787. PMID 24124323
- [Background] Bredenoord AJ, Weusten BL, Curvers WL, Timmer R, Smout AJ. Determinants of perception of heartburn and regurgitation. Gut. 2006 Mar;55(3):313-8. doi: 10.1136/gut.2005.074690. Epub 2005 Aug 24. PMID 16120760
- [Background] Holten KB, Wetherington A, Bankston L. Diagnosing the patient with abdominal pain and altered bowel habits: is it irritable bowel syndrome? Am Fam Physician. 2003 May 15;67(10):2157-62. PMID 12776965
- [Background] Kay L, Jorgensen T, Jensen KH. The epidemiology of irritable bowel syndrome in a random population: prevalence, incidence, natural history and risk factors. J Intern Med. 1994 Jul;236(1):23-30. doi: 10.1111/j.1365-2796.1994.tb01115.x. PMID 8021568
- [Background] Yao X, Yang Y, Zhang S, Shi Y, Zhang Q, Wang Y. The impact of overlapping functional dyspepsia, belching disorders and functional heartburn on anxiety, depression and quality of life of Chinese patients with irritable bowel syndrome. BMC Gastroenterol. 2020 Jul 6;20(1):209. doi: 10.1186/s12876-020-01357-1. PMID 32631285
- [Background] Talley NJ, Dennis EH, Schettler-Duncan VA, Lacy BE, Olden KW, Crowell MD. Overlapping upper and lower gastrointestinal symptoms in irritable bowel syndrome patients with constipation or diarrhea. Am J Gastroenterol. 2003 Nov;98(11):2454-9. doi: 10.1111/j.1572-0241.2003.07699.x. PMID 14638348
- [Background] Hachem C, Shaheen NJ. Diagnosis and Management of Functional Heartburn. Am J Gastroenterol. 2016 Jan;111(1):53-61; quiz 62. doi: 10.1038/ajg.2015.376. Epub 2016 Jan 5. PMID 26729546
- [Background] Schuster MM. Defining and diagnosing irritable bowel syndrome. Am J Manag Care. 2001 Jul;7(8 Suppl):S246-51. PMID 11474909